CLINICAL TRIAL: NCT05577299
Title: Factors Affecting Brown Adipose Tissue (BAT) Activation in Cancer Patients Undergoing 18F-FDG-PET/CT
Brief Title: Factors Affecting BAT Activation in PET/CT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Nabil Helbawi, resident doctor, Assiut University
Other Study IDs: BAT activation in PET/CT
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Factors Affecting BAT Activation in PET/CT
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET/CT — 18F-fluorodeoxyglucose positron emission tomography/computed tomography (18FFDG PET/CT) is a non-invasive imaging modality used for staging and surveillance of various types of malignancies through imaging of glucose metabolism in cancer cells.

SUMMARY:
The aim of the present study is to evaluate the factors affecting BAT activation in 18F-FDG-PET/CT in different tumours

DETAILED DESCRIPTION:
Positron emission tomography (PET)/CT with fluorine-18 fluorodeoxyglucose (18F-FDG) is currently a standard diagnostic tool for identifying tumours and their metastases as well as infectious or inflammatory lesions.1-3 High physiological uptake of 18F-FDG is found in organs with high glucose metabolism, such as the brain and heart. One particular tissue with high 18F-FDG uptake that can interfere with scan interpretation is brown fat.4 Brown fat, or brown adipose tissue (BAT), is involved in non-shivering thermogenesis and creates heat through glucose metabolism. It is found mostly in the cervical, supraclavicular and thoracic paravertebral regions,5 and some is also found in the axillae, mediastinum and abdomen.6 Although it is usually simple for nuclear medicine physicians to recognize BAT uptake through its typical pattern and from the low attenuation in the CT scan, high uptake in BAT can still be mistaken for a malignant lesion or cause false-negative results by obscuring small metastases and decrease diagnostic confidence of the scan professional reading. BAT has a preferential distribution over the body and a preferential occurrence in female, younger and thinner patients. It mainly interferes with scan interpretation in tumours that occurs at younger age and is located in or metastasize to the head, neck and peri clavicular/axillary regions, such as melanoma of the upper body, breast cancer, and head and neck cancers, but it can also cause problems in lung and other cancers.7.8

ELIGIBILITY:
Inclusion Criteria:

* This study will include all patients presented with different types of tumors.
* patients conscious to provide informed consent

Exclusion Criteria:

* • Patients who have contraindications to PET/CT scanning such as: a blood glucose level higher than 150-200 mg/dL, uncontrolled diabetics.

  * Intolerance of PET/CT due to claustrophobia will be excluded from the study.
  * Patients under age of 18

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cancer patients undergoing PET/CT
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
the main factors that affect appearance of BAT in PET/CT studies and try to avoid these factors. | from 7/2019 to 7/2022
  the amount and SUV max of the detected BAT activation in PET scan correlated with the patient prognosis.